CLINICAL TRIAL: NCT05926089
Title: Acute Phase Reactant in Non-COVID-19 Community Acquired Pneumonia
Brief Title: Acute Phase Reactant in Non-COVID-19 Bacterial Pneumonia
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Kamal Ibrahim Hassan, Assistant Professor of pulmonology, Cairo University
Other Study IDs: MS-358-2020
Record Dates: First submitted 2023-06-28; First posted 2023-07-03 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Pneumonia; Acute-Phase Reaction
MeSH Terms: conditions — Pneumonia; Acute-Phase Reaction | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — • Complete blood picture, differential leucocytic count and platelets count: Done by The newly developed automated hematology analyzer (Sysmex, Kobe, Japan) enumerates and classifies blood cells by a combination of direct current detection and flow cytometry. (Daves et al., 2015).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood sampling — blood sampling to measure APR

SUMMARY:
This study is a cross-sectional study, was conducted at Chest department of Kasr Al-ainy Hospital, Cairo university during the period between October 2020 and April 2021.

The aim of the work was to evaluate levels of acute phase reactants(APR) in Non-COVID-19 bacterial pneumonia, and to correlate between levels of APR and the disease severity.

DETAILED DESCRIPTION:
51 patients were included in our study, diagnosed as Non-COVID pneumonia

Inclusion criteria:

1. PCR(polymerase chain reaction) negative for COVID.
2. All patients of both sexes with pneumonia .

Exclusion criteria:

1. Non pulmonary infections.
2. Post surgery patients.
3. Renal patients.
4. hepatic patients.
5. Cardiac patients.
6. Recent pulmonary embolism.

Methodology in details:

All patients were subjected to:

1. Full history with emphasis on:

   * Epidemiological features (age, gender).
   * Risk factors (smoking, DM).
   * Clinical presentation (cough, Fever and duration of illness).
2. Clinical examination (local chest examination).
3. Laboratory investigations: venous blood samples were taken to measure APR

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 negative bacterial pneumonia

Exclusion Criteria:

* COVID-19 positive
* other non-pulmonary infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients( 51 patients diagnosed as non-COVID19 Pneumonia) were subjected to:
  1. Full historywith emphasis on:
     * Epidemiological features .
     * Risk factors (smoking, DM).
     * Clinical presentation (cough, Fever and duration of ilness).
  2. Clinical examination (local chest examination).
  3. Laboratory investigations: venous blood samples were taken for:• Complete blood picture, differential leucocytic count and platelets count, ESR ,CRP, d-dimer and ferritin
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
measurement of APR levels in non-Covid-19 pneumonia | 6 months
  assessment of the level of APR and its relation to disease severity

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy school of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No